CLINICAL TRIAL: NCT04191720
Title: A Randomized Control Trial to Assess the Impact of Weighted Blankets on Anxiety Among Inpatients With Anorexia Nervosa and Avoidant Restrictive Food Intake Disorder: a Study Protocol
Brief Title: Assessing the Impact of Weighted Blankets on Anxiety Among Inpatients With Anorexia Nervosa: a Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Rachel Ohene, Occupational Therapist, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-0596
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Anorexia Nervosa; Avoidant/Restrictive Food Intake Disorder; Anxiety
Keywords: anorexia nervosa; weighted blankets; occupational therapy; anxiety; deep pressure stimulation; randomized control trial
MeSH Terms: conditions — Anorexia Nervosa; Avoidant Restrictive Food Intake Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group, or usual care group, will receive occupational therapy standard of care. Occupational therapy standard of care provide training, education, and therapeutic activities including relaxation strategies. These coping mechanisms are aimed at reducing the impact of anxiety on a patient's performance and participation in necessary and meaningful activities of daily living, refeeding and medical stabilization. Specifically, these interventions will include diaphragmatic and yogic breathing exercises, mindfulness-based cognitive therapy (MBCT) education and exercises, therapeutic restorative yoga activities, occupational therapy group participation, aromatherapy, identifying and promoting engagement in meaningful leisure activities, client-centered sensory diets to provide patients with consistent preferred sensory experiences, and individualized checklists and schedules to grade the self-initiation of effective coping strategies.
- Weighted blanket group (Experimental): In the weighted blanket intervention group, patients will receive usual occupational therapy care in addition to a weighted blanket. The patient will be given an appropriately weighted blanket, within 1 lb +/- of 10% of body weight as measured on day of admission. Further, the occupational therapy will provide education to the patient on the use of the weighted blanket. Patients will be free to use the weighted blanket at their discretion, however, during meals, over the shoulders or head, and during ambulation, weighted blanket use will not be permitted.
  Interventions: Other: Weighted blanket

INTERVENTIONS:
Other: Weighted blanket — Patients that were randomly assigned to the intervention group received a weighted blanket to use at their will to reduce anxiety
  Arms: Weighted blanket group

SUMMARY:
The aim of this study is to conduct a randomized control trial (RCT) to assess the efficacy of weighted blankets (WB), on anxiety for patients with severe anorexia nervosa (AN) and avoidant restrictive food intake disorder (ARFID) in an inpatient medical setting. We hypothesize that using weighted blankets will reduce anxiety in these patient populations.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) has one of the highest mortality rates of any psychiatric disorder with anxiety being a common comorbidity. The standard of care for inpatient medical stabilization for patients diagnosed with AN is a multidisciplinary approach with emphasis on nutrition, psychotherapy, and medical management of complaints. Weighted blankets, an example of deep pressure stimulation, have been shown to reduce anxiety. However, not much is known about the effect of weighted blankets in the eating disorder population. Therefore, this randomized control trial (RCT) protocol outlines a study design for assessing the effect of weighted blankets on patients with AN.

A two-arm RCT design will be implemented for this study. A convenience sample of 24 patients will be enrolled with 12 patients in the control and intervention groups based on inclusion criteria. The control group will receive Denver Health's standard of care for patients admitted to its well-known medical stabilization unit for patients with extreme form of eating disorders, while the intervention group will receive both the standard of care and a weighted blanket. A mixed-design ANOVA will be performed to explore differences in the Beck's Anxiety Inventory and Subjective Units of Distress Scale between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with AN-R, AN-BP, or ARFID upon admission (per Diagnostic and Statistical Manual-V criteria)
* Moderate/Major Anxiety per initial evaluation score using BAI
* OT assessment

Exclusion Criteria:

* Pregnant or nursing mothers

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Anxiety reduction | BAI measured during OT evaluation and through study completion, an average of 1 year
  Beck Anxiety Inventory (BAI)
Anxiety reduction | SUDS are measured during OT evaluation and through study completion, an average of 3 weeks
  Subjective Units of Distress Scale (SUDS)

SECONDARY OUTCOMES:
Times weighted blankets are used | Behaviors will be documented every 2 hours over the course of treatment, through study completion, an average of 3 weeks
  Ratio of times weighted blankets were used vs when not in use

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ohene, MOT, Principal Investigator — Denver Health Hospital and Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
If we decide to share the data, we would ask researchers to reach out to the PI

REFERENCES:
- [Background] Hoek HW. Incidence, prevalence and mortality of anorexia nervosa and other eating disorders. Curr Opin Psychiatry. 2006 Jul;19(4):389-94. doi: 10.1097/01.yco.0000228759.95237.78. PMID 16721169
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Khalsa SS, Portnoff LC, McCurdy-McKinnon D, Feusner JD. What happens after treatment? A systematic review of relapse, remission, and recovery in anorexia nervosa. J Eat Disord. 2017 Jun 14;5:20. doi: 10.1186/s40337-017-0145-3. eCollection 2017. PMID 28630708
- [Background] Paslakis G, Maas S, Gebhardt B, Mayr A, Rauh M, Erim Y. Prospective, randomized, double-blind, placebo-controlled phase IIa clinical trial on the effects of an estrogen-progestin combination as add-on to inpatient psychotherapy in adult female patients suffering from anorexia nervosa. BMC Psychiatry. 2018 Apr 10;18(1):93. doi: 10.1186/s12888-018-1683-1. PMID 29631553
- [Background] Nakai Y, Nin K, Noma S, Teramukai S, Wonderlich SA. Characteristics of Avoidant/Restrictive Food Intake Disorder in a Cohort of Adult Patients. Eur Eat Disord Rev. 2016 Nov;24(6):528-530. doi: 10.1002/erv.2476. Epub 2016 Sep 4. PMID 27594387
- [Background] Elliot ML. Figured world of eating disorders: occupations of illness. Can J Occup Ther. 2012 Feb;79(1):15-22. doi: 10.2182/cjot.2012.79.1.3. PMID 22439288
- [Background] Chakraborty K, Basu D. Management of anorexia and bulimia nervosa: An evidence-based review. Indian J Psychiatry. 2010 Apr;52(2):174-86. doi: 10.4103/0019-5545.64596. PMID 20838508
- [Background] Sebastian MR, Wiemann CM, Hergenroeder AC. Rate of weight gain as a predictor of readmission in adolescents with eating disorders. Int J Adolesc Med Health. 2019 Feb 26;33(4). doi: 10.1515/ijamh-2018-0228. PMID 30807289
- [Background] Altman SE, Shankman SA. What is the association between obsessive-compulsive disorder and eating disorders? Clin Psychol Rev. 2009 Nov;29(7):638-46. doi: 10.1016/j.cpr.2009.08.001. Epub 2009 Aug 16. PMID 19744759
- [Background] Nicely TA, Lane-Loney S, Masciulli E, Hollenbeak CS, Ornstein RM. Prevalence and characteristics of avoidant/restrictive food intake disorder in a cohort of young patients in day treatment for eating disorders. J Eat Disord. 2014 Aug 2;2(1):21. doi: 10.1186/s40337-014-0021-3. eCollection 2014. PMID 25165558
- [Background] Meier SM, Bulik CM, Thornton LM, Mattheisen M, Mortensen PB, Petersen L. Diagnosed Anxiety Disorders and the Risk of Subsequent Anorexia Nervosa: A Danish Population Register Study. Eur Eat Disord Rev. 2015 Nov;23(6):524-30. doi: 10.1002/erv.2402. Epub 2015 Sep 8. PMID 26347124
- [Background] Chen H-Y, Yang H, Chi H-J. Physiological Effects of Deep Touch Pressure on Anxiety Alleviation: The Weighted Blanket Approach. Journal of Medical and Biological Engineering. 2013;33(5):463-70.
- [Background] Edelson SM, Edelson MG, Kerr DC, Grandin T. Behavioral and physiological effects of deep pressure on children with autism: a pilot study evaluating the efficacy of Grandin's Hug Machine. Am J Occup Ther. 1999 Mar-Apr;53(2):145-52. doi: 10.5014/ajot.53.2.145. PMID 10200837
- [Background] Grandin T. Calming effects of deep touch pressure in patients with autistic disorder, college students, and animals. J Child Adolesc Psychopharmacol. 1992 Spring;2(1):63-72. doi: 10.1089/cap.1992.2.63. PMID 19630623
- [Background] Krauss KE. The effects of deep pressure touch on anxiety. Am J Occup Ther. 1987 Jun;41(6):366-73. doi: 10.5014/ajot.41.6.366. PMID 3688151
- [Background] Reynolds S, Lane SJ, Mullen B. Effects of deep pressure stimulation on physiological arousal. Am J Occup Ther. 2015 May-Jun;69(3):6903350010p1-5. doi: 10.5014/ajot.2015.015560. PMID 25871605
- [Background] Kimball JG, Lynch KM, Stewart KC, Williams NE, Thomas MA, Atwood KD. Using salivary cortisol to measure the effects of a Wilbarger protocol-based procedure on sympathetic arousal: a pilot study. Am J Occup Ther. 2007 Jul-Aug;61(4):406-13. doi: 10.5014/ajot.61.4.406. PMID 17685173
- [Background] Sylvia LG, Shesler LW, Peckham AD, Grandin T, Kahn DA. Adjunctive deep touch pressure for comorbid anxiety in bipolar disorder: mediated by control of sensory input? J Psychiatr Pract. 2014 Jan;20(1):71-7. doi: 10.1097/01.pra.0000442942.01479.ce. PMID 24419314
- [Background] VandenBerg NL. The use of a weighted vest to increase on-task behavior in children with attention difficulties. Am J Occup Ther. 2001 Nov-Dec;55(6):621-8. doi: 10.5014/ajot.55.6.621. PMID 12959226
- [Background] Champagne T, Stromberg N. Sensory approaches in inpatient psychiatric settings: innovative alternatives to seclusion & restraint. J Psychosoc Nurs Ment Health Serv. 2004 Sep;42(9):34-44. doi: 10.3928/02793695-20040901-06. PMID 15493494
- [Background] Chen HY, Yang H, Meng LF, Chan PS, Yang CY, Chen HM. Effect of deep pressure input on parasympathetic system in patients with wisdom tooth surgery. J Formos Med Assoc. 2016 Oct;115(10):853-859. doi: 10.1016/j.jfma.2016.07.008. Epub 2016 Aug 24. PMID 27568389
- [Background] Tanner BA. Validity of global physical and emotional SUDS. Appl Psychophysiol Biofeedback. 2012 Mar;37(1):31-4. doi: 10.1007/s10484-011-9174-x. PMID 22038278